CLINICAL TRIAL: NCT06064630
Title: The Effect of Telemedicine-Based APAP Management on 24-Hour Ambulatory Blood Pressure in Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaosong Dong, Clinical Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022PHB359-001
Record Dates: First submitted 2023-08-22; First posted 2023-10-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine treatment group (Other): Telemedicine group need to complete sleep-related questionnaires online. Participants in the telemedicine group will learn Home sleep apnea testing(HSAT) online and then complete overnight monitoring at home. Patients diagnosed with OSA after HSAT monitoring will receive standardized APAP treatment. At 1 month of APAP treatment, participants in the telemedicine group will be followed up by phone/video to check their APAP treatment compliance. After 3 months of APAP treatment, the telemedicine group will be followed up by phone/video to check their APAP treatment compliance at 3 month, and they will finish 24-hour ambulatory blood pressure monitoring.
  Interventions: Device: Automatic continuous positive airway pressure
- Outpatient treatment group (Other): Outpatient group need to complete sleep-related paper questionnaires at sleep center. The sleep technicians will explain to the patients how to use the Home sleep apnea testing (HSAT) and then they will complete overnight monitoring at home. Patients diagnosed with OSA after HSAT monitoring will receive standardized APAP treatment. At 1 month of APAP treatment, participants in the outpatient group will be followed up at sleep center to check their APAP treatment compliance. After 3 months of APAP treatment, the outpatient group will be followed up to check their APAP treatment compliance at 3 month, and they will finish 24-hour ambulatory blood pressure monitoring.
  Interventions: Device: Automatic continuous positive airway pressure

INTERVENTIONS:
Device: Automatic continuous positive airway pressure — Automatic continuous positive airway pressure (APAP) is the routine and first line treatment for patients with sleep apnea

SUMMARY:
Epidemiological studies have shown that OSA is closely related to the occurrence and development of cardiovascular diseases, especially hypertension. At present, there are 66 million patients with moderate to severe OSA in China, and the current diagnosis and treatment of OSA is mainly completed in the sleep center of the hospital, which is time-consuming and laborious, resulting in the delayed diagnosis and treatment of a large number of patients, making about 80% of potential OSA patients have not been diagnosed and treated in time. With the development of the Internet technologies, telemedicine has been increasingly applied to the diagnosis, treatment and management of chronic diseases with its advantages of convenience, interactivity, efficiency, sharing, coherence and breaking through the limitations of time and space. Our center has initially built a remote diagnosis and treatment management model for OSA. Compared with the traditional medical model, the medical and health economic analysis shows that the OSA diagnosis and treatment model based on telemedicine is more cost-effective, but its clinical efficacy needs to be further verified. Hypertension is a common complication in OSA patients, and continuous positive airway pressure (PAP) has a significant hypertensive effect in the treatment of OSA. However, whether clinical management based on remote diagnosis and treatment mode can achieve the same therapeutic effect as traditional face-to-face diagnosis and treatment mode in improving ambulate blood pressure in OSA patients needs to be further clarified. This study will compare the improvement of 24 hour ambulatory blood pressure in patients under the Telemedicine-Based APAP Management and the traditional outpatient management through a single-center randomized controlled trial.

DETAILED DESCRIPTION:
Patients presenting with snoring were randomized to telemedicine-based or conventional outpatient management. We compared changes in 24-hour ambulatory blood pressure after 3 months of APAP therapy between groups. Secondary outcomes included treatment adherence, patient-reported symptoms and biological parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected OSA and recommended to sleep center for HSAT monitoring;
2. Voluntary and signed informed consent;
3. Access to the Internet, email and phone calls;
4. Lived in Beijing for the last three months (subjects randomly assigned to the outpatient treatment group were able to travel to and from the sleep center);
5. Fluent Chinese expression;

Exclusion Criteria:

1. Blood pressure cuff should not be used (e.g., circumference of upper arm > 55cm, history of breast cancer, structural lesions of upper limb);
2. Has been treated with a CPAP or oral appliance;
3. Cardiac insufficiency, NYHA classes III-IV;
4. Clear central sleep apnea (AHI≥15 times/hour, central events > 50%);
5. Expected life span < 2 years;
6. Pregnant women;
7. History of kidney failure or kidney transplantation;
8. Attention deficit hyperactivity disorder, use of wakefulness drugs;
9. Less than 5 hours of sleep per night on weekdays combined with other sleep problems (e.g., shift work, night shift, circadian rhythm disturbance);
10. Oxygen is needed when awake or sleeping;
11. Unstable condition: unstable angina pectoris, uncontrolled hypertension, severe COPD, tumor progression, or unstable mental illness;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
24-hour ambulatory blood pressure | 12weeks
  24-hour mean blood pressure(Primary), Daytime mean blood pressure, Nighttime mean blood pressure, 24-hour Systolic blood pressure (SBP), Daytime SBP, Nighttime SBP, 24-hour Diastolic blood pressure (DBP), Daytime DBP, Nighttime DBP.

SECONDARY OUTCOMES:
The compliance of APAP treatment | 12weeks
  Evaluate the use time of auto positive airway pressure therapy per night, including the proportion of the number of days with good compliance and the average daily use of the daily use of the APAP during treatment.
Sleepiness symptom | 12weeks
  Daytime sleepiness was measured by the Epworth Sleepiness Scale (ESS, score range 0-24), with higher scores indicating greater sleepiness
Sleep Functional Outcome | 12weeks
  Disease-specific functional status was assessed using the 10-item Functional Outcomes of Sleep Questionnaire (FOSQ-10), a validated instrument designed to quantify the impact of sleepiness on daytime functioning. The FOSQ-10 comprises 10 items, yielding a total score ranging from 5 to 20, with higher scores indicating better daytime functional status and less impairment in daily activities.
OSA-specific quality of life | 12 weeks
  OSA-specific quality of life was evaluated with the 32-item Quebec Sleep Questionnaire (QSQ), which measures five domains (daytime sleepiness, diurnal symptoms, nocturnal symptoms, emotions, and social interactions) on a 7-point Likert scale, with higher scores indicating better quality of life.
Sleep quality | 12 weeks
  General sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI). The global PSQI score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Mood and depressive symptoms | 12 weeks
  Mood and depressive symptoms were assessed using the 10-item Center for Epidemiologic Studies Depression Scale (CES-D-10), a self-report questionnaire evaluating the frequency of depressive symptoms over the past week. Each item is rated on a 4-point scale (0-3), yielding a total score of 0-30, with higher scores indicating greater depressive symptom burden.
Insomnia symptoms | 12 weeks
  Insomnia symptoms were assessed using the Insomnia Severity Index (ISI). The total ISI score ranges from 0 to 28, with higher scores indicating more severe insomnia.

OTHER OUTCOMES:
Liver enzyme | 12 weeks
  Serum liver enzyme levels including alanine aminotransferase (ALT) and aspartate aminotransferase (AST) will be measured as indicators of hepatic function. These enzymes are routinely quantified in fasting blood samples using standardized biochemical assays. ALT and AST elevations reflect hepatocellular injury, inflammation, or metabolic stress. Tests will be performed by the hospital's central biochemical laboratory. ALT and AST values will be reported in international units per liter (U/L)
Lipid profile | 12 weeks
  The lipid profile includes measurements of fasting total cholesterol (TC), triglycerides (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C). These markers are measured in the hospital's biochemical laboratory and are established indicators of lipid metabolism and cardiovascular risk. Results will be expressed in mmol/L according to laboratory standards.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaosong Dong, Principal Investigator — Sleep Medicine Center, Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No